CLINICAL TRIAL: NCT06106737
Title: A Modified Calculation Formula for Meibomian Gland Grading
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20231020
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-10

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- previous calculation formula
- modified calculation formula

SUMMARY:
The meibomian gland (MG) is a modified sebaceous gland located in the upper and lower eyelids. The grades of MG loss (i.e. meiboscore) is calculated as the ratio between the area of the MGs and the eyelids, and this calculation is based on the two-dimensional digital infrared images.In the current formula, the area of the eyelid is the denominator. However, because the eyelids need to be flipped over for the examination and evaluation, and there may be interobserver variability in the measurement of the area of the eyelids. Aging and involutional eyelid disorders, such as ptosis, ectropion, and entropion, may lead to laxity or deformation of eyelids, and impact the shape and area of eyelid area consequently.These factors could cause inaccuracy in current evaluation method, and impact the grading and evaluation of treatment efficacy of MGD, especially in self-controlled studies, such as in clinical trials.

In this study, the investigators propose to use a modified calculation formula for the grading of MGs. The investigators could measure the white to white (WTW) distance of cornea, and then calculate the area of cornea (i.e. corneal base area) accordingly.Unlike the eyelid, the WTW distance does not change significantly during aging or between sexes.Thus, the investigators hypothesize that using the corneal base area as the new denominator in the formula for the grading of MG loss is a better way comparing with the conventional method.

ELIGIBILITY:
Inclusion Criteria:

* people aged 18 to 80

Exclusion Criteria:

* Exclusion criteria included contact lens wearer, history of eye surgeries, systemic health conditions affecting ocular health and those who were unable to cooperate with examinations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient population
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
the area of the MGs and the whole eyelids | Baseline (Once a subject has enrolled in research)
the WTW distance of the cornea | Baseline (Once a subject has enrolled in research)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China